CLINICAL TRIAL: NCT03392922
Title: A Comparison the Intubation of a Left Sided Double Lumen Tube and the Uniblocker Under the Guidence of Chest Computed Tomography Image
Brief Title: A Comparison the Intubation of a Left Sided Double Lumen Tube and Uniblocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 966168
Record Dates: First submitted 2017-12-16; First posted 2018-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2017-12

CONDITIONS: Therapeutic Procedural Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uniblocker (Experimental): The BBs have more advantages than DLT: easier insertion especially in patients with difficult airway18 and no need to exchange the tube when mechanical ventilation is required after surgery
  Interventions: Device: Uniblocker
- Left-sided Double-lumen Tube (Experimental): the double-lumen tube (DLT) is the most commonly used device for OLV
  Interventions: Device: Left-sided Double-lumen Tube

INTERVENTIONS:
Device: Uniblocker — The BBs have more advantages than DLT: easier insertion especially in patients with difficult airway18 and no need to exchange the tube when mechanical ventilation is required after surgery.
  Arms: Uniblocker
Device: Left-sided Double-lumen Tube — the double-lumen tube (DLT) is the most commonly used device for OLV
  Arms: Left-sided Double-lumen Tube

SUMMARY:
One-lung ventilation (OLV) is required for the most thoracic surgery to facilitate surgical visualization by collapsing the lung. The double-lumen tube (DLT) and Uniblocker are the commonly used device for OLV.The objective of our study was to comparison the safety and effectiveness of the intubation of the Left-sided Double-lumen Tube and the Uniblocker under the guidence of chest computed tomography (CT) image.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is required for the most thoracic surgery to facilitate surgical visualization by collapsing the lung. The double-lumen tube (DLT) and Bronchial blockers (BBs) are the commonly used device for OLV.The objective of this study is to comparison the safety and effectiveness of the intubation of the Left-sided Double-lumen Tube and the Uniblocker under the guidence of chest computed tomography (CT) image(the operator count the number of CT slices (slice thickness is 5mm) from vocal cord slice to carina slice to calculate the distance between vocal cord and carina) then measure a distance on the DLT or Uniblocker from the upper edge of the cuff to the mouth side and made a marker on the DLT or Uniblocker.During the intubation the operator insert the DLT or Uniblocker into the trachea via video laryngoscope, after passing the glottis the DLT or Uniblocker are advanced toward the left main-stem bronchus, once the anesthesiologist see the marker on the DLT or the Uniblocker just above the vocal cord stop the insertion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing left side thoracic surgery

Exclusion Criteria:

* 1.Age>70 or <18 years 2.ASA classifications >III 3.BMI >35kg/m2 4.Modified Mallampati classification ≥III 5.Thoracic surgery within the last one month 6.Severe cardiopulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
The incidence of the optimal position on the first attempt | 1 year
The incidence of the injuries of bronchi and carina. | 1 year

SECONDARY OUTCOMES:
The time for the intubation of Uniblocker or Left-sided Double-lumen Tube | 1 year
The incidence of lung adequacy collapse | 1 year
The incidence of Uniblocker displacement | 1 year
The incidence of sore throat and hoarseness postoperative | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Derived] Liu Z, Zhao L, Zhu Y, Bao L, Jia QQ, Yang XC, Liang SJ. The efficacy and adverse effects of the Uniblocker and left-side double-lumen tube for one-lung ventilation under the guidance of chest CT. Exp Ther Med. 2020 Apr;19(4):2751-2756. doi: 10.3892/etm.2020.8492. Epub 2020 Feb 5. PMID 32256757